CLINICAL TRIAL: NCT02048345
Title: Gastrointestinal Behavior of Posaconazol in Healthy Volunteers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Bart Hens, Pharmacist, KU Leuven
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: DDD13POSA
Record Dates: First submitted 2013-06-23; First posted 2014-01-29 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: Healthy
Keywords: ten mL suspension of posaconazol (Noxafil) together with 240mL water will be taken by the volunteer in a fasted state; ten mL suspension of posaconazol (Noxafil) together with 240mL water will be taken by the volunteer in a fed state; two point six mL of suspension that is dissolved in 247mL water will be administered to the volunteer by the stomach catheter in a fasted state; two point six mL of suspension that is dissolved in 247mL water will be administered to the volunteer by the stomach catheter in a fed state

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Suspension, fasted state (Experimental): Suspension Noxafil will be administered in the fasted state to the volunteers.
  Interventions: Drug: Suspension Fasted State
- Suspension, with sugar (delay gastric emptying) (Experimental): Suspension will be co-administered with glucose to delay the gastric emptying time
  Interventions: Drug: Suspension Fed State
- Solution, fasted state (Experimental): A solution (by acidifying the suspension in water to pH 1.2) will be administered to healthy volunteers in a fasted state.
  Interventions: Drug: Solution Fasted State
- Solution, with sugar (delaying gastric emptying) (Experimental): A solution of posaconazol (by acidifying the suspension in water to pH 1.2) will be administered together with sugar to delay the gastric emptying.
  Interventions: Drug: Solution Fed State

INTERVENTIONS:
Drug: Suspension Fasted State
  Arms: Suspension, fasted state
Drug: Suspension Fed State
  Arms: Suspension, with sugar (delay gastric emptying)
Drug: Solution Fasted State
  Arms: Solution, fasted state
Drug: Solution Fed State
  Arms: Solution, with sugar (delaying gastric emptying)

SUMMARY:
The aim of this study is to understand the behavior of posaconazol gives as a suspension and solution in the gastrointestinal tract in human volunteers. The investigators know that supersaturation for this compound can be achieved by the influence of the gastrointestinal tract: The acid environment of the stomach creates a optimized environment for the basic compound to reach a high solubility, while the neutral environment of the small intestine creates a low solubility environment for the compound. The transit from stomach to small intestine gives the opportunity for the drug to create a supersaturated solution. Giving the drug as a solution to the healthy volunteer makes sure that precipitation is not occurring in the stomach and that precipitation has to happen in the small intestine. After all, supersaturation is a state that is not thermodynamic stable and always will want to precipitate. Giving the drug as a suspension to the healthy volunteers, can make it possible that still some particles of the drug are not in dissolution and that those particles will flow to the small intestine where other particles easily can bind to. This will make that almost the whole supersaturated solution is immediately precipitated.

The investigators want to give the suspension by the authorized drug called Noxafil. On the other hand an aqueous solution will be made by adjusting the pH to 1.2 (which is conform with the pH of the stomach) and given to the volunteers by the stomach catheter. This 2 formulations will be tested in a fasted state and a fed state (by giving 2 Ensure plus shakes to the volunteers before the experiment starts). After intake of the formulation, gastric and duodenal fluids will be aspirated by the catheters and analyzed at their laboratory. So the four conditions the investigators want to study are:

1. 10 mL Suspension of posaconazol (Noxafil 40mg/mL) together with a glass of 240 mL water in a fasted state
2. 250 mL solution of posaconazol, by dissolving 2.6 mL autohorized suspension (Noxafil) in 247 mL water, adjusted to pH 1.2 by hydrochloric acid given to the volunteer in a fasted state.
3. 10 mL Suspension of posaconazol (Noxafil 40mg/mL) together with a glass of 240 mL water in a fed state (by giving 20 minute before intake of the formulation, 2 ensure plus shakes)
4. 250 mL solution of posaconazol, by dissolving 2.6 mL autohorized suspension (Noxafil) in 247 mL water, adjusted to pH 1.2 by hydrochloric acid given to the volunteer in a fed state (by giving 20 minute before intake of the formulation, 2 ensure plus shakes).

By getting more knowledge about the behavior of posaconazol (interplay supersaturation / precipitation) more insights can be achieved for the development of supersaturating drug delivery systems.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years Healthy volunteers

Exclusion Criteria:

* disease Hiv, Hepatitis B, Hepatitis C Pregnant Drug abuse

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Concentration-time profile in stomach and small intestine for posaconazol | These concentrations will be measured for 4 hours, together by taking blood samples to see how the drug will be transported to the blood circulation (PK profile for 48 hours)

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven Gasthuisberg, Leuven, Belgium